CLINICAL TRIAL: NCT00703001
Title: Waukesha Smiles: Dental Outreach to Low-income Waukesha Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Kenneth G. Schellhase, MD; Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2007I-45
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1--Educational Intervention (Active Comparator): Students in this arm will receive several in-class educational modules on basic oral health topics.
  Interventions: Behavioral: Educational Intervention
- 2--Referral intervention (Active Comparator): Parents of student subjects will receive assistance in accessing oral health care for their child
  Interventions: Behavioral: Referral Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — students in this arm will receive several oral health educational modules in class
  Arms: 1--Educational Intervention
Behavioral: Referral Intervention — Parents of enrolled children will receive assistance in accessing oral health care for their child
  Arms: 2--Referral intervention

SUMMARY:
The Waukesha Smiles Project will compare approaches to improve oral health habits and increase access to basic dental care for low-income children in Waukesha, Wisconsin through a school-based outreach program of oral health promotion, screening and referral.

DETAILED DESCRIPTION:
A. HYPOTHESIS / SPECIFIC AIMS: The purpose of Waukesha Smiles: Dental Outreach to Low-income Children will be to improve oral health habits and increase access to primary and preventive dental care for low-income children in the city of Waukesha.

The typical forms of dental decay seen in children, also called dental "caries," are the result of a transmissible infectious disease process that is enabled by poor oral hygiene and dietary choices.1-5 When unchecked, this process leads to pain and tooth loss, which can in turn lead to disfigurement, self-esteem problems, impaired nutrition, and even systemic disease.3, 6 Access to basic dental care and good oral health habits can reduce preventable dental disease and these associated outcomes.7 However, poor oral health habits are more prevalent among children from lower socioeconomic strata.7-9 And limited access to primary/preventive dental care is common for low income and/or minority children, and represents a major health risk for these specific populations.9, 10 Self-pay for care is a major barrier for low-income families.9, 10 Children with Title 19-related dental insurance (Medicaid) also face similar barriers from limited provider acceptance of this program: due to low levels of reimbursement many dentists in the Waukesha area limit the number of Title-19 patients in their practices, and some do not accept this insurance at all.10, 11 Furthermore, adequate access to dental care alone is not sufficient to assure oral health: regular dental visits cannot compensate for poor oral health habits.

The Waukesha County Dental Clinic (WCDC) will open in January 2008 with a mission to serve low-income uninsured and underinsured county residents. This new clinic will serve a critical function in our community. However, despite the increased access to care that the Waukesha County Dental Clinic will provide, we expect that many eligible low-income Waukesha children will still not receive needed dental care for a variety of reasons. These include: lack of awareness of the clinic; persistent concern about financial burdens; lack of understanding about the benefits of routine dental care; logistical barriers; and language and cultural barriers. Moreover, we expect that if basic oral health habits could be improved in Waukesha children, the need for anything but preventive dental care would diminish.

We hypothesize that an Educational Intervention, consisting of brief monthly classroom presentations on oral health plus monthly distribution of a new toothbrush and tooth paste, will lead to improved oral health outcomes among low-income 3rd grade students when compared to a Referral Intervention wherein children will receive a detailed referral and assistance finding a dentist after an oral health screening exam. Our primary outcomes are rates of untreated dental caries, and the proportion of children needing early or urgent dental care.

B. DESIGN/ METHODS: Aim/Objective 1: Assemble a cohesive study team, including parent advisory board and bilingual study staff for oral health outreach interventions.

Aim/Objective 2: Develop and prepare Educational and Referral Interventions Aim/Objective 3: Conduct both interventions in two phases, using a cross-over approach so that all children in the study receive both interventions.

Aim/Objective 4: Evaluate, sustain, and disseminate this partnership for child oral health improvement.

Waukesha Smiles will compare two different school-based strategies for improving oral health among 400 3rd grade children in 9 different elementary schools in the city of Waukesha with high proportions of low-income students. All students will receive screening oral health exams at the beginning and end of each intervention; parents will be provided with the exam results and recommendations for care. Intervention groups will divided by school, so that all children in the same school receive the same intervention (as close to 200 children per group as feasible). However, to maximize community benefit from this project and allay concerns about participation in research, we will use a crossover design such that the schools will swap interventions after the first 12 months (Phase I). Thus Intervention Phase II will provide the same interventions for the same duration in the opposite schools, again with pre- and post-intervention oral screening exams.

INTERVENTION PHASE I, First Cohort: Participants in the Referral Intervention arm will receive a specific referral for dental care as indicated by their baseline exam; detailed information about the Waukesha County Dental Clinic (WCDC), a new clinic opening to serve uninsured and low-income county residents; and reminders and active follow-up by study staff to assist children and parents in overcoming barriers to accessing recommended care. INTERVENTION PHASE I, Second Cohort:The Educational Intervention arm will consist of monthly classroom visits by a dental education team (dental hygienist plus assistant) to provide brief oral health education modules, and to distribute a new toothbrush and new tube of toothpaste each month. On the first visit, participants will be given a timer to promote proper brushing duration. In INTERVENTION PHASE II, the first and second cohorts will swap interventions, allowing all children in the study to receive both interventions.

C. VARIABLES (predictor / outcome; stopping rules / endpoint)

D. STATISTICS: We will use McNemar's test and other basic statistical testing methods to determine if the results of the pre- and post-intervention oral health assessment exams are significantly different in terms of the prevalence of our primary outcomes: untreated caries and the need for early/urgent dental care. Because our groups are not randomized, in order to directly compare differences in outcomes between interventions (Referral vs. Education) we will construct a logistic regression model to allow adjustment for multiple baseline differences between groups; variables in the model will include school attended, low-income status, and parental education level. Using descriptive statistics we will also analyze (a) parental surveys for changes in oral health knowledge/attitude/behavior, and changes in perceived barriers to dental care, (b) rates of follow-through on recommended dental care, and (c) rates of Emergency Department visits at two local hospitals for pediatric dental problems with patient zip codes lying in our schools' catchment area. We will not seek to track Emergency visits by patient name. Family Medicine residents' experiences with the project will be evaluated through their rotations. Lastly, through feedback given to the study team, community partners, and investigators, we will seek to determine the feasibility of sustaining one or both of these interventions in Waukesha schools, and to determine how best to disseminate our results to others.

E. RISKS: We believe the risks in this study are relatively minimal, and will include:

1. possible embarrassment of the child due to identification of dental needs during oral health assessment
2. unable to receive recommended dental care despite assistance with referrals, availability of new clinic catering to low-income and Medicaid patients, etc.
3. transmission of infection during oral health assessment
4. breech of confidentiality

F. BENEFITS: This project will expand on and sustain the success of a 2004 HWPP planning grant ("Creating a Community-Academic Partnership to Improve the Oral Health of Waukesha County"). This ongoing partnership led to the development of the Waukesha County Dental Clinic to address unmet oral health needs. This success is evidence of a productive working relationship and long-term commitment of financial and professional resources from each partner according to their particular strengths. This productive partnership will continue to meet at least biweekly during this project, and demonstrates commitment and ability to attain the elements of the Community-Academic Partnership Model such as realistic assessment of needs/barriers, ability to garner broad support, shared passion for improving oral health, creating and attaining measurable goals, mutual trust, and sharing resources.

We will measure the impact of this project through several key outcomes. At the end of the each intervention period, we will analyze interval differences in the oral health screening exam results for each study arm; specific attention will be paid to differences between groups in rates of untreated caries, appearance of new interval lesions, and regression of early lesions. We will measure the proportion of children requiring early or urgent dental care. We will also track the outcomes of referrals to the WCDC, and pediatric Emergency Department visits for acute dental problems at local hospitals using zip code methods. To maximize the health impact of this project, we will develop a how-to manual and resource guide of best practices that will allow other Wisconsin communities to take this program "off the shelf." In addition, family medicine residents will take lessons learned back to the underserved areas where they tend to practice.

ELIGIBILITY:
Inclusion Criteria:

* 3rd grade student (school year 2007-2008) in one of 9 selected Waukesha School District schools serving a population with high poverty rates

Exclusion Criteria:

* cognitive delay that would prohibit student from giving meaningful assent to participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Improved oral health status of subjects as measured by caries index | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Schellhase, MD MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States